CLINICAL TRIAL: NCT07029334
Title: Effectiveness Evaluation in the SHINE Research Programme - Social Prescribing for Adults and Elderly: The Path to Effective Implementation
Brief Title: Effectiveness Evaluation of Social Prescribing
Status: Recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Volunteer Center Sydhavnen (Unknown); GP cluster Vesterbro-Sydhavnen (Unknown)
Responsible Party: Principal Investigator, Ove Andersen, Professor, MD, PhD, Hvidovre University Hospital
Other Study IDs: P-2024-17318
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Loneliness; Health Related Quality of Life
Keywords: Social Prescribing; Public Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SP participants: Participants in the intervention who has provided consent to participate in the effectiveness evaluation.
  Interventions: Other: Social Prescribing
- SP participants - controls (registry data): Matched controls (registry data) 1:4 selected from the same GP clinics and matched to cases based on age group, gender, and Charlson Comorbidity Index score.

INTERVENTIONS:
Other: Social Prescribing — The SP intervention consists of a series of intervention components delivered across the SP pathways:
  Intervention components
  GP:
  1. Social prescribing from physician to patient
     Link Worker:
  2. Initial phone contact
  3. Clarification and follow-up consultations
  4. Personalized matching with local services and activities
  5. Care coordination
  6. Introductory visits to local services and activities
  7. Accompanied (if needed)
  8. Follow-up conversations
  9. Concluding conversations
  10. Group-based courses
      GP / Link Worker:
  11. Re-prescribing (where appropriate)
  Each intervention component is described in detail in the TIDieR checklist
  Groups: SP participants

SUMMARY:
Social Prescribing (SP), or Social Henvisning (SH) in Denmark, integrates healthcare with social and cultural services to address social determinants of health. The 'Social Prescribing Vesterbro-Sydhavnen' initiative, launched in fall 2024 as part of usual care, aims to involve general practitioners (GP) as primary prescribers to social services through a dedicated link worker, enhancing early intervention and connecting healthcare with community support.

This evaluation aims to assess the effectiveness of the 'Social Prescribing Vesterbro-Sydhavnen' project as part of the Implementation Research Programme SHINE.

The primary outcomes are: changes in contacts with general practice, unplanned hospital contacts and emergency calls (1813) as well as change in patients' perception of loneliness and health-related Quality of life.

DETAILED DESCRIPTION:
Social Prescribing (SP), or Social Henvisning (SH) in Denmark, integrates healthcare with social and cultural services to address social determinants of health. Internationally, SP improves patient well-being, reduces loneliness, and lowers healthcare utilization. Countries like the United Kingdom, Canada, and Australia have shown its effectiveness in reducing hospital admissions and supporting vulnerable populations.

The 'Social Prescribing Vesterbro-Sydhavnen' initiative, launched in fall 2024 as part of usual care, aims to involve general practitioners (GP) as primary prescribers to social services through a dedicated link worker, enhancing early intervention and connecting healthcare with community support.

This evaluation aims to assess the effectiveness of the 'Social Prescribing Vesterbro-Sydhavnen' project, in the following named as SP-intervention.

Information about the experimental group The participants in this evaluation are all patients participating in the SP intervention upon referral from their GP. The investigators anticipate that up to 500 patients from around 15 GPs in 10 clinics will participate in the SP-intervention, hereof a sample of 315 in the analysis of this evaluation. Participants are recruited consecutively in the GP clinics starting from summer 2025.

The target group of the SP-intervention are adults (+18) with or at risk of complex health and social challenges or with a high level of both elective and acute visits to general practice, including socially related consultations.

Research questions:

Research question 1: How does the SP intervention impact healthcare service utilization for the participating patients?

Research question 2: How does the SP intervention impact the perceived degree of loneliness and quality of life in participating patients?

All outcomes in this evaluation are presented both as a total and stratified by each GP clinic, age-group, gender, education, employment, civil status, and migration background.

Other secondary research questions:

What are the demographic and clinical characteristics of citizens utilizing the SP project, including their baseline levels of perceived loneliness and quality of life?

What characterizes the clinics that refer patients to the SP intervention? Descriptive statistics on General Practitioners regarding the clinic characteristics and population affiliated with the clinic:

* Number of patients per clinic
* Number of patients per GP
* Age distribution
* Gender distribution
* Socioeconomic distribution
* Disease burden distribution (Charlson Comorbidity Index Score, Dual Diagnosis, Triple Diagnosis)
* Type of clinic

The study will also explore the following research questions related to impact and influencing factors of the SP Intervention:

* Are the effects of the SP intervention influenced by participants' socio-economic background, pre-existing health conditions, or other variables?
* How do different types of services in the SP intervention compare in terms of their effect on participants' well-being, loneliness, and healthcare utilization over time?
* How do the frequency and duration of engagement in the SP project influence its effects on healthcare utilization and well-being?
* What factors lead to dropouts of the SP-intervention?

Project design:

This effectiveness evaluation is designed as a quasi-experimental, prospective cohort study with a real-world approach, following a per-protocol analysis. The evaluation outcomes feeds into the Implementation Programme SHINE which employs a Hybrid Type II Effectiveness-Implementation Design.

The participants in this evaluation are all patients participating in the SP intervention upon referral from their GP. Participants are recruited consecutively in the GP clinics starting in June, 2025.

The target group of the SP-intervention are adults (+18) with or at risk of complex health and social challenges or with a high level of both elective and acute visits to general practice, including socially related consultations.

Data sources:

Research Question 1 is analysed using Danish national registry data without requiring informed consent. A case-control design is applied, where cases include all patients prescribed the SP intervention by their GP in the Vesterbro-Sydhavnen area of Copenhagen. Controls are selected from the same GP clinics and matched to cases based on age group, gender, and Charlson Comorbidity Index score.

Research Question 2 is analysed using patient-reported outcomes collected after obtaining informed consent from SP intervention participants. This analysis does not include a control group.

Recruitment and informed consent After being prescribed to participate in the SP intervention by their GP, patients have an initial meeting with the link worker (in Danish: Brobygger). During this visit, the link worker introduces the evaluation, provides participant information, and explains the evaluation process in detail. Participation is voluntary. Patients who wish to consider their participation further are given a two-week reflection period and may bring a relative to a follow-up meeting before deciding.

If they agree to participate, they provide informed consent digitally on a tablet. Consent forms and responses are securely uploaded to REDCap, a GDPR-compliant data capture system hosted by the Capital Region of Denmark. Data is stored securely, and only authorized project staff have access. Participants can withdraw their consent at any time without consequences for their future treatment.

Data collection:

Following consent, the link worker or designated project staff administers Patient Reported Outcome (PRO) questionnaires, assessing Health-Related Quality of Life (HRQoL) and loneliness, on a tablet. The PRO data after 3 and 9 months is collected by a link to REDCap sent to the participants by SMS message or email. In the event of participant dropout, the link worker or other project staff will attempt to collect PRO data at the time of dropout.

If participants do not respond to the 3- or 9-month follow-up via SMS or email, project staff will follow up by telephone to attempt contact. Registry data will be retrieved after the final patient has completed the 9-month assessment - see data sources in detail below.

Data sources:

The description of the baseline profile and assess outcome measures, this evaluation uses registry data from Statistics Denmark, the Register of Healthcare Providers, the National Health Insurance Service Register, the National Prescription Registry, the Danish National Patient Register (LPR), and the Danish Register of Causes of Death, utilizing the Personal Identification Number (CPR) on all SP-intervention participants provided by the GPs/brobygger.

Statistical considerations:

Baseline characteristics of participants and controls will be summarized using means (SD) or medians (IQR) for continuous variables and frequencies (%) for categorical variables.

Primary Analysis - Healthcare Utilization Outcomes Unadjusted rates of GP contacts, unplanned hospital contacts, and emergency calls (1813) will be calculated for intervention and control groups.

Multivariable Poisson or negative binomial regression models will estimate rate ratios (RRs) for changes in healthcare contacts, adjusting for age and other relevant covariates (e.g. education).

Changes in medication prescriptions will be compared between intervention and control group (assessed by dosage/number of prescriptions 6 months prior and 9 months after intervention).

Primary Analysis - Patient-Reported Outcomes (Loneliness & HRQoL) Changes in loneliness (T-ILS and De Jong Gierveld Loneliness Scale) and HRQoL (EQ-5D-5L and EQ-VAS) from baseline to 3 and 9 months follow-up will be analysed using linear mixed-effect models, adjusting for baseline scores and covariates (e.g. age, use of psychotropic medication and civil status).

Secondary Analysis Participation and non-attendance in the SP intervention will be modelled using logistic regression, including demographic and clinical factors.

Other analysis

All primary analyses will be stratified by GP clinic (stratification analysis) Alternative definitions of multimorbidity (e.g., number of chronic conditions, dual diagnosis, triple diagnosis vs. Charlson Comorbidity Index) (sensitivity analysis)

Interactions between mental health and socioeconomic status to explore effect modification of intervention and control group. (interaction/sub analysis).

If missing data can be assumed to be missing at random, multiple imputation will be used to account for missing data.

Sample size:

The power calculation is based on the outcome measures of change in GP visits. Since GP visit rates for the study population under investigation are unknown, the investigators have based the calculation on the GP rate from a UK study with a similar intervention, which reported a median annual rate of 8.3. This is rescaled to 9 months, equalling a rate of 6.225 visits per 9 months (Carnes m.fl. 2017). With a power of 0.8, a significance level of 0.05, and a minimal rate reduction of 10%, a sample of 315 cases is required. To account for confounder adjustments, additional cases are included, resulting in a final sample of 350 cases.

Ethics:

This non-interventional evaluation of usual care in the primary healthcare sector, integrates data from Danish registers with participant-reported information collected through questionnaires administered at three time points over the course of the SP intervention. The investigators do not consider this study to pose any harm or cause discomfort to the participants.

The project will adhere to the ethical guidelines set by the Danish Council for Independent Research. The data collected will be stored and processed in accordance with the Danish Data Protection Agency and the EU General Data Protection Regulation and registered in the records of the Capital Region of Denmark. The investigators will obtain written informed consent from all participants following approval and recommendations from the Regional Research Ethics Committee.

The study will be conducted adhering to the ethical principles of the Helsinki Declaration, ensuring ethically responsible research, including informed consent, protection of participants' rights, risk assessment, and transparency in the study's purpose and methodology. Additionally, the project is registered with the Capital Region of Denmark's data registry P-2024-17318.

ELIGIBILITY:
All participants in the SP intervention are invited consecutively to participate in the effectiveness evaluation by the Link Worker. There are no exclusion or inclusion criteria in the effectiveness evaluation of the SP intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GP´s work with the following inclusion and exclusion criteria when detecting eligible patients for the SP-intervention:
  INCLUSION CRITERIA
  * Citizens aged 18+
  * In need of social support that can complement treatment in general practice or disease prevention
  * Motivated or can be motivated to participate.
  * Can be contacted via phone or email.
  * Reside in Vesterbro-Sydhavnen, Copenhagen Municipality
  EXCLUSION CRITERIA
  * Severe mental illness, other serious disabilities, or substance abuse that prevents the patient from participating in voluntary or municipal services.
  * Lack of basic language skills in Danish or English, which corresponds to levels A1-A2 of the Common European Framework of Reference for Languages (CEFR), indicating that the individual has very limited or no proficiency in the language.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate ratios for change in contacts with GP | From the date the Link Worker received the social prescription to 3 and 9 months thereafter.
  Primary Outcome:
  • Change in contacts with general practice (all type of contacts)
Rate ratios for change in unplanned hospital contacts | From the date the Link Worker received the social prescription to 3 and 9 months thereafter.
  Primary Outcome:
  • Change in unplanned hospital contacts
Rate ratios for change in emergency calls (1813) | From the date the Link Worker received the social prescription to 3 and 9 months thereafter.
  Primary Outcome:
  • Change in emergency calls (1813)
Change in the perceived degree of loneliness assessed by T-ILS | From the enrollment date to 3 and 9 months after the Link Worker has received the social prescription.
  Primary Outcome:
  • Change in perception of loneliness - assessed by Three-Item Loneliness Scale (T-ILS).
  The scale uses three response categories: Hardly ever = score 1, Some of the time = score 2, Often = score 3. Higher scores means worse outcome.
Change in the perceived degree of loneliness - assessed by De Jong Gierveld Loneliness Scale | From the enrollment date to 3 and 9 months after the Link Worker has received the social prescription.
  Primary Outcome:
  • Change in perception of loneliness - assessed by De Jong Gierveld Loneliness Scale
  On the positively worded items, the neutral and negative answers are scored as "1" (Yes=0, More or less=1, and No=1). A higher score means a worse outcome.
Change in quality of life - assessed by EQ-5D-5L | From the enrollment date to 3 and 9 months after the Link Worker has received the social prescription.
  Primary Outcome:
  • Change in perception of Health-related Quality of Life (HRQoL) - assessed by EQ-5D-5L. The EQ-5D-5L instrument covers five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with five response levels: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems, 5 = extreme problems; higher scores indicate worse outcomes. Dimension-level responses are aggregated into a single utility index using the Danish value set (range < 0 [health states worse than death] to 1 [full health]); lower index scores reflect poorer health.
Change in quality of life - assessed by EQ-VAS (visual analog scale) | From the enrollment date to 3 and 9 months after the Link Worker has received the social prescription.
  Primary Outcome:
  • Change in perception of Health-related Quality of Life (HRQoL) - assessed by EQ-VAS (visual analog scale).
  Tthe minimum value = 0 and maximum value = 100. A higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change in prescribed medication use (rate and dosage) | 6 months prior and 9 months after the date the Link Worker received the social prescription
  Change in medication prescriptions (e.g., prescriptions for psychotropic drugs and pain medication) will be compared between intervention and control group (assessed by dosis/number of prescriptions

OTHER OUTCOMES:
Participation in the Social Prescribing intervention. | Assessed 3 and 9 months after the link worker has received the SP referral from the GP
  Frequency of participation in services (I am there every time, I am there most of the time, I am there sometimes, I am there almost never, I have not been there yet)
Service types in Social Prescribing | End of followup: 9 months after the link worker has received the SP referral from the GP
  Categorical classification of services participants are referred to
Dropout of evaluation | End of followup: 9 months after the link worker has received the SP referral from the GP
  Categorical classification of reasons for discontinuation in the evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, Professor, MD, Principal Investigator — Department of Clinical Research, Copenhagen University Hospital, Hvidovre; Jeanette Wassar Kirk, PhD, Associate Professor, Study Chair — Department of Clinical Research, Copenhagen University Hospital, Hvidovre
Locations (1):
- Volunteer Center Sydhavnen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from Statistics Denmark but restrictions apply to the availability of these data, which were used under licence for the current study, and therefore they are not publicly available.

REFERENCES:
- [Derived] Kirk JW, Oldrup LS, Lindstrom MB, Hansen JA, Broholm-Holst M, Andersen O. SHINE - social prescribing for adults and the elderly: the path to effective implementation. A study protocol. Implement Sci Commun. 2025 Oct 14;6(1):104. doi: 10.1186/s43058-025-00791-0. PMID 41088466
- See also: Link to the paper used for the sample size calculation based on GP visit rates — https://doi.org/10.1186/s12913-017-2778-y